CLINICAL TRIAL: NCT04550806
Title: The Predictive Ability of Glycated Albumin Combined With Body Composition for Gestational Diabetes Mellitus Diagnosis
Brief Title: Glycated Albumin Combined With Body Composition for Gestational Diabetes Mellitus Prediction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-1703
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM
- non-GDM

SUMMARY:
This study is going to investigate the predictive ability of glycated albumin combined with body composition, including body weight, BMI, fat free mass and fat mass for gestational diabetes mellitus (GDM) diagnosis.

DETAILED DESCRIPTION:
The prevalence of GDM is increasing all over the world. It has bad influence for both pregnant women and fetus. Early treatment is useful for GDM prevention. Therefore early screening is important for healthcare doctors to detect the potential patients. Glycated albumin (GA) is an optimal index for blood glucose evaluation compared to HbA1c, however it may be influenced by body weight and composition. The investigators are going to investigate the predictive ability of glycated albumin combined with body composition, including body weight, BMI, fat free mass and fat mass for gestational diabetes mellitus (GDM) diagnosis. This study recruit pregnant women before 12 weeks of their pregnant age and test GA level and body composition via bioelectrical impedance analysis. During 24-28 weeks of pregnant age, all participants will do the glucose tolerant test for GDM diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-45
* Healthy, without heart disease, liver or kidney dysfunction, immune system or metabolic or infectious disease,

Exclusion Criteria:

* Diabetes that appeared before pregnancy
* Pregnant with medical disease, such as asthma, hypertension, cardiovascular diseases, kidney diseases or liver disease.
* Hormone use in the recent 1 year
* Assisted reproduction pregnancy
* Multiple births
* Cannot complete the blood test or body composition examination

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women at first trimester
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of GA combined with body composition for GDM diagnosis | May 2021
  prediction ability of GA and body compostion

SECONDARY OUTCOMES:
correlative factors for GDM | May 2021
  regression model to detect correlative factors for GDM
GDM prediction model establishment | May 2021
  multiple regression model to establish screening system for GDM

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, MD, Study Director — Clinical nutrition department of Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
we can update the information collected of this study